CLINICAL TRIAL: NCT03233568
Title: Use of Indirect Calorimetry in Dietary Setting in Obese Subjects: Retrospective Observational Study
Brief Title: Use of Indirect Calorimetry in Obesity
Status: Completed | Type: Observational
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Anna Ferrulli, Sub-Investigator, Ospedale San Donato
Other Study IDs: CALO/Obesity
Record Dates: First submitted 2017-07-21; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Metabolism Disorder; Overweight and Obesity
MeSH Terms: conditions — Metabolic Diseases; Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Indirect Calorimetry group (IC group): Group who performed indirect calorimetry. REE measured by indirect calorimetry.
  Interventions: Diagnostic Test: Indirect calorimetry
- NO Indirect Calorimetry group (NO-IC group): Group who did not perform indirect calorimetry. Resting Energy Expenditure calculated by Harris-Benedict formula

INTERVENTIONS:
Diagnostic Test: Indirect calorimetry — Indirect calorimetry will be performed by using an open-circuit calorimeter (Sensor Medics, Italy). Indirect calorimetry is the reference method for energy expenditure determination. A canopy hood covered the patient's head and expired air is extracted by a pump to be analyzed by metabolic cart sensors; flow rate is directly measured with a digital turbine flowmeter. After an overnight fast, patients will asked to lay supine in complete physical rest, not sleeping or talking for approximately 20-25 minutes, at a room temperature ranged between 22 and 24°C. The mean REE for each participant considers the last 15-20 minutes of measurements corresponding to steady state.
  Software of calorimeter will be set for minute-by-minute reading report of VO2 (Oxygen flow) and VCO2 (Carbon dioxide flow) measurement.
  Parameters obtained by Indirect Calorimetry will be the Resting Energy Expenditure and the Respiratory Quotient (RQ)
  Groups: Indirect Calorimetry group (IC group)

SUMMARY:
The investigators will retrospectively analyze and compare data of 2 groups of overweight and obese patients: subjects who followed a diet based on Resting Energy Expenditure (REE) measured by indirect calorimetry and subjects who followed a diet based on REE estimated by the Harris-Benedict equation. Propensity score adjustment will be used to adjust for known differences between the 2 groups

ELIGIBILITY:
Inclusion Criteria:

* BMI >25
* Age ranging from 20 to 86 years

Exclusion Criteria:

* BMI<25
* Age <20
* Age >86

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To collect clinical data of a total population comprising patients referred to our Endocrinology-Diabetes Outpatient Clinic, in the period from April 2012 through October 2016.
  In this retrospective study, will be considered patients with an age ranging from 20 to 86 years, with overweight (25 ≤ BMI ≤ 29.9) or obesity (BMI ≥ 30), requiring dietary intervention for weight control.
  Statistical analysis will perform on overweight and obese patients divided into two subgroups: IC group and NO-IC group.
  Anthropometric status and metabolic biomarkers will re-evaluated at check-ups performed after 3 months, 6 months, 12 months and 18 months from the baseline.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Weight in Indirect Calorimetry group and in NO Indirect Calorimetry group | 18 months
  To compare body weight variation (kg) in two groups of overweight or obese patients: subjects who followed a diet formulated on REE measured by IC (IC group) and subjects who followed a diet based on REE predicted by the Harris-Benedict formula (NO-IC group)
BMI in Indirect Calorimetry group and in NO Indirect Calorimetry | 18 months
  To compare BMI variation (kg/m^2) in two groups of overweight or obese patients: subjects who followed a diet formulated on REE measured by IC (IC group) and subjects who followed a diet based on REE predicted by the Harris-Benedict formula (NO-IC group)

SECONDARY OUTCOMES:
Weight in male/female in Indirect Calorimetry group and in NO indirect Calorimetry group | 18 months
  To identify gender differences in weight variation (kg) between IC and NO-IC groups
BMI in male/female in Indirect Calorimetry group and in NO indirect | 18 months
  To identify gender differences in BMI variation (kg/m^2) between IC and NO-IC groups

OTHER OUTCOMES:
Weight in adequate to predicted REE and in NOT adequate to predicted REE subpopulations | 18 months
  to compare body weight variation (kg) in two sub-populations of the IC-group: subjects with adequate to predicted REE and subjects with not adequate to predicted REE
BMI in adequate to predicted REE and in NOT adequate to predicted REE subpopulations | 18 months
  to compare BMI variation in two sub-populations of the IC-group: subjects with adequate to predicted REE and subjects with not adequate to predicted REE
Weight in subjects with RQ<0.9 and subjects with RQ>0.9 | 18 months
  to compare body weight variation in 2 subpopulation of the IC group: subjects with an RQ ≤ 0.9 and subjects with RQ > 0.9.
BMI in subjects with RQ<0.9 and subjects with RQ>0.9 | 18 months
  BMI variation in 2 subpopulation of the IC group: subjects with an RQ ≤ 0.9 and subjects with RQ > 0.9.
Glucose in Indirect Calorimetry group and in NO Indirect Calorimetry Group | 18 months
  to identify differences in glucose (mg/dl) variation between IC and NO-IC groups
Tryglycerides in Indirect Calorimetry group and in NO Indirect Calorimetry Group | 18 months
  to identify differences in tryglycerides (mg/dl) variation between IC and NO-IC groups
Total cholesterol (mg/dl) in Indirect Calorimetry group and in NO Indirect Calorimetry Group | 18 months
  to identify differences in cholesterol variation between IC and NO-IC groups
Hemoglobin in Indirect Calorimetry group and in NO Indirect Calorimetry Group | 18 months
  to identify differences in glycated hemoglobin (%) variation between IC and NO-IC groups
Uric acid in Indirect Calorimetry group and in NO Indirect Calorimetry Group | 18 months
  to identify differences in uric acid (mg/dl) variation between IC and NO-IC groups

CONTACTS AND LOCATIONS:
Overall Officials: Livio Luzi, Professor, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- San Donato Hospital, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Massarini S, Ferrulli A, Ambrogi F, Macri C, Terruzzi I, Benedini S, Luzi L. Routine resting energy expenditure measurement increases effectiveness of dietary intervention in obesity. Acta Diabetol. 2018 Jan;55(1):75-85. doi: 10.1007/s00592-017-1064-0. Epub 2017 Nov 3. PMID 29101542